CLINICAL TRIAL: NCT06925230
Title: Arthroscopic Assisted Volar, Dorsal or Combined Capsulodesis in Scapholunate Ligament Injury
Acronym: case series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD 61/2023
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Scapholunate Interosseous Ligament Injury; SLLI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- arthroscopic assisted volar scapholunate capsulodesis (Other): arthroscopic assisted combined volar capsulodesis using PDS 2.00 sutures
  Interventions: Procedure: arthroscopic assisted volar scapholunate capsulodesis; Procedure: arthroscopic assisted dorsal scapholunate capsulodesis; Procedure: arthroscopic assisted combined volar and dorsal scapholunate capsulodesis

INTERVENTIONS:
Procedure: arthroscopic assisted volar scapholunate capsulodesis — arthroscopic assisted volar scapholunate capsulodesis using PDS 2.00 sutures
  Other Names: volar scapholunate capsuloligamentodesis
Procedure: arthroscopic assisted dorsal scapholunate capsulodesis — arthroscopic assisted dorsal scapholunate capsulodesis using PDS 2.00 sutures
Procedure: arthroscopic assisted combined volar and dorsal scapholunate capsulodesis — arthroscopic assisted combined volar and dorsal scapholunate capsulodesis using PDS 2.00 sutures

SUMMARY:
The aim of this case series study is to test the efficacy of arthroscopic assisted volar, dorsal or combined scapholunate capsulodesis in the management of scapholunate ligament injuries.

DETAILED DESCRIPTION:
The aim of this case series study is to test the efficacy of arthroscopic assisted volar, dorsal or combined scapholunate capsulodesis in the management of scapholunate ligament injuries. All patients will be assessed preoperatively by careful history taking , full general and local examination and radiological evaluation using wrist plain X-rays (Standard PA, clenched-fist PA , PA in ulnar deviation , lateral projection in neutral ,flexion and extension ) and wrist Magnetic resonance imaging.an informed written consent was taken before any surgery. The procedure starts with a standard radiocarpal and then midcarpal arthroscopy. During the arthroscopic examination ,several factors are assessed, including the location of the SLIL injury (volar, membranous, dorsal, or complete), the condition of the cartilage, the reducibility of the carpus, and other associated pathologies like TFCC injury. Classification is done using Geissler Classification, Garcia Elias Classification and EWAS classification.Volar capsulodesis using Hayman Lui et al or Del Pinal et al method and/or dorsal capsulodesis using original Mathoulin technique or combined capsulodesis were done.

ELIGIBILITY:
Inclusion Criteria:

* Sex: both sexes.
* Age: above 18 years
* Lesion: subacute or chronic scapholunate ligament injury
* partial and complete SLIL tears

Exclusion Criteria:

* Acute scapholunate ligament injury
* irreducible carpal malalignment
* posttraumatic arthritis
* associated fractures that could affect the functional outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
wrist range of motion | preoperative and postoperative after 3months , 6months , 9months and 12months
  wrist range of motion degrees in flexion , extension, radial deviation and ulnar deviation.

SECONDARY OUTCOMES:
scapholunate gap | preoperative and postoperative scapholunate gaps after 3months , 6months , 9months and 12months
  scapholunate gap in PA wrist plain Xray is the distance between middle of scaphoid and middle of lunate bones in PA wrist plain Xray in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt